CLINICAL TRIAL: NCT06485310
Title: Interest of a TEteleconsultation of a Psychological Support Nurse on Psychological Distress in Patients With a Primary Malignancy of the Central Nervous System Between the Announcement of the Diagnosis and the First Treatment
Brief Title: Interest of a TEteleconsultation of a Psychological Support Nurse on Psychological Distress in Patients With a Primary Malignancy of the Central Nervous System
Acronym: TECAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/CHU/02
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Cancer; Psychological Distress
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELECONSULTATION (Experimental): Teleconsultation with a nurse for psychological support, after the diagnosis has been announced, before hospitalization for the first treatment (chemotherapy, surgery, radiotherapy) in addition to the standard practice.
  Interventions: Other: Teleconsultation for psychological support
- NO TELECONSULTATION (No Intervention): The control group will be cared for according to standard practice (without teleconsultation)

INTERVENTIONS:
Other: Teleconsultation for psychological support — Teleconsultation with a nurse for psychological support, after the diagnosis has been announced, before hospitalization for the first treatment (chemotherapy, surgery, radiotherapy) in addition to the standard practice
  Arms: TELECONSULTATION

SUMMARY:
The goal of this clinal trial is to compare the effectiveness of nurse-led teleconsultation with usual care (intervention group) on psychological distress in patients with primary malignant tumors of the central nervous system between diagnosis and first anti-cancer treatment, versus usual care alone (control group).

Participants will be randomized into two groups :

* group A) intervention: usual care + nurse teleconsultation for psychological support
* group B) control: usual care alone

Enrolment = Day0 (D0)

Participants will :

* groups A and B: D0: complete 4 questionnaires (Quality of Life, Screening for Distress, Screening for Anxiety and Depression, Social Support Questionnaire)
* Group A : D0+2/4 das : nursing teleconsultation for psychological support
* Groups A and B: D0+10days : telephone call to complete the same 4 questionnaires as at inclusion
* Group A : D0+15days: semi-directive interview, at home, for voluntary patients.

DETAILED DESCRIPTION:
The expected benefits are as follows:

For the patient :

* Reduction in pre-treatment psychological distress
* Reduced pre-treatment anxiety and depression
* Better understanding of disease and treatments
* Better adherence to the care proposed in the treatment pathway
* Reduced stress during first hospital treatment

For healthcare professionals :

* Early detection of psychological distress
* Early detection of unmet needs and appropriate individualized responses
* Establishment of a climate of trust between patient and caregiver
* Improved professional practices

For the healthcare system :

* Lower healthcare costs (fewer anxiolytic treatments, etc.)
* Therapy to be integrated into the treatment pathway of patients with central nervous system cancer
* Reduced socio-territorial inequalities in healthcare provision

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over
* being treated for a primary malignant tumor of the central nervous system (positive biopsy)
* with a Mini-Mental State score greater than 24
* not receiving first-line treatment (chemotherapy, targeted radiotherapy, surgery)
* with a distress score above 3 on the Psychological Distress Thermometer
* have access to computer equipment equipped with a microphone and webcam (smartphone, computer)
* able to read, write and speak French
* have given free and informed consent
* being affiliated to a social security scheme

Exclusion Criteria:

* with a history of psychiatric illness
* with recurrent cancer of the cerebral nervous system
* having begun first-line treatment (drug therapy, curative surgery, radiotherapy or palliative care)
* under guardianship, curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Distress thermometer | 10 days
  Comparison of the change in psychological distress score, measured using the psychological distress screening tool (from National Comprehensive Cancer Network) between the 2 groups between inclusion (T0) and before the first anti-cancer therapy (T1).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Reunion Island - Neurosurgery department, Saint-Pierre-des-Corps, Reunion, France

IPD SHARING:
Plan to Share IPD: No